CLINICAL TRIAL: NCT06942351
Title: Effect of Walnuts on Cognitive Function and Gut Microbiome in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon State University (Other)
Collaborators: California Walnut Commission (Other)
Responsible Party: Principal Investigator, Emily Ho, Endowed Chair and Director, Linus Pauling Institute University Distinguished Professor, College of Health, Oregon State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: LPI-1153
Record Dates: First submitted 2025-04-08; First posted 2025-04-24 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-04

CONDITIONS: Aging; Inflammation Biomarkers
Keywords: gut microbiome; walnuts; cognitive function

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study staff performing cognitive tests and analyzing samples and cognitive data will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walnuts (Active Comparator): Daily consumption of 1.5 ounces (42.5 g) of plain walnuts for 12 weeks
  Interventions: Other: Walnuts
- Crackers (Placebo Comparator): Daily consumption of non-whole grain crackers for 12 weeks (caloric equivalent to 1.5 ounces of plain walnuts)
  Interventions: Other: Crackers

INTERVENTIONS:
Other: Walnuts — Daily consumption of 1.5 ounces of plain walnuts for 12 weeks
  Arms: Walnuts
Other: Crackers — Daily consumption of non-whole grain crackers for 12 weeks (caloric equivalent to 1.5 ounces of plain walnuts)
  Arms: Crackers

SUMMARY:
The purpose of this study is to examine the impact of daily consumption of walnuts for 12 weeks on cognitive function, markers of inflammation and oxidative stress, and the gut microbiome in healthy adults age 55 years and older.

DETAILED DESCRIPTION:
The investigators will determine the extent to which daily consumption of walnuts by older adults for 12 weeks influences cognitive function and whether improvements are associated with changes in the resident gut microbiota. The investigators propose that age-related cognitive decline can be mitigated by consuming walnuts, by modulating the microbiota and microbial metabolites and decreasing oxidative stress and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years or older
* Able to hear well enough to understand spoken instructions and questions
* Able to see well enough to read and respond to printed instructions and fill out questionnaires (corrective lenses are allowed)
* Able to write legibly and move a computer joystick with at least one hand (i.e., no injury or connective tissue or joint disorder that would impair ability to write or make hand movements)
* Able to speak, read, and understand English
* Score of greater than 79 on water maze learning task
* Willing to maintain current eating patterns
* Willing and able to complete the cognitive tests
* Willing to stop consuming almonds, Brazil nuts, cashews, chestnuts, hazelnuts, macadamia nuts, peanuts, pecans, pistachios, walnuts, persimmons and pomegranates for 14 weeks. - are nuts or contain ellagitannins or ellagic acid - compounds/foods of interest for this study
* Willing to limit oak aged wines and spirits to 1 serving/day and limit blackberries (including similar berries like boysenberries, marionberries, and olallieberries), cloudberries, cranberries, currants, elderberries, lingonberries, raspberries, strawberries, wolfberries, other native berries; guava, mango, muscadine grapes, nectarines, peaches, plums, pluots to 1 cup/day for 14 weeks; REMAIN CONSISTENT (consistent intake levels of): Coffee, tea, apple, apricots, blueberries, cherries, grapes (table/common)
* Willing to stop probiotic supplements 2 weeks prior to and during the study (14 weeks)

Exclusion Criteria:

* Consumption of walnuts, pecans, and chestnuts combined greater than 2 oz / week in the past 3 months.
* Use of oral antibiotics in the past month
* Regular use of oral anti-inflammatory medications in the past month
* Nut, wheat, or gluten allergy/intolerance
* Pregnant or planning to become pregnant during the study period
* Weighs less than 110 pounds
* Diagnosis of sickle cell disease
* Susceptibility to motion sickness
* Consumes 3 or more alcoholic drinks daily
* History of smoking tobacco products, including e-cigarettes and vaporizers in the past 2 years (smokeless tobacco use not exclusionary)
* Use of psilocybin or cannabis products (including CBD-only products) in the past 2 years
* Current treatment for alcohol or other substance use disorder
* History of heart attack, heart failure, or stroke, including transient ischemic attack
* History of liver disease or kidney disease requiring dialysis
* History of cancer in the past 5 years (Skin cancer that was only surgically treated is not exclusionary)
* History of bariatric surgery (e.g., gastric bypass, gastric banding, sleeve gastrectomy, etc.) or disorders (e.g., Crohn's disease, unmanaged celiac disease, ulcerative colitis)
* History of thyroid disorder that requires medication, but subject is not taking medication
* History of chronic bronchitis or emphysema
* Diagnosis of dementia or Alzheimer's disease
* History of head injury requiring hospitalization or loss of consciousness > 5 minutes
* History of chronic migraines (for at least 3 months, headache occurring on 15 or more days per month, where at least 8 of those headache days have migraine symptoms)
* Blood pressure above 159 (systolic) or 99 (diastolic) mm Hg
* Corrected vision worse than 20/50
* Score of less than 10/15 on Ishihara color vision test or diagnosis of color blindness
* Score of less than 26/30 on Mini-Mental State Exam
* Score of greater than 15 on Center for Epidemiologic Depression survey
* History of disease or disorder which causes cognitive impairment, including but limited to: attention-deficit/hyperactivity disorder (ADHD), amyotrophic lateral sclerosis, autism, bipolar disorder, Down's syndrome, encephalitis, epilepsy/seizures, human immunodeficiency virus (HIV), Huntington's disease, Korsakoff's psychosis, multiple sclerosis, Parkinson's disease, or psychotic disorders (e.g., schizophrenia, schizoaffective disorder, schizophreniform disorder)
* Current and regular use of any of the following medications: insulin, opioids, anti-seizure medications, psychotropic medications: stimulants, anti-psychotics, or medications that cause daytime drowsiness or difficulty concentrating

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Cognitive function - memory | 0 and 12 weeks
  Change from baseline at week 12: age adjusted standard scores (higher score reflects positive outcome)
Cognitive function - memory | 0 and 12 weeks
  Change from baseline at week 12: proximity (lower score reflects positive outcome)
Cognitive function - cognitive flexibility | 0 and 12 weeks
  Change from baseline at week 12: age adjusted standard scores (higher score reflects positive outcome)
Cognitive function - cognitive flexibility | 0 and 12 weeks
  Change from baseline at week 12: proximity (lower score reflects positive outcome)
Cognitive function - speed of processing | 0 and 12 weeks
  Change from baseline at week 12: age adjusted standard scores (higher score reflects positive outcome)
Gut microbiome composition | 0 and 12 weeks
  Change from baseline at week 12: microbiome composition
Lipid oxidation levels | 0 and 12 weeks
  Change from baseline at week 12: plasma malondialdehyde (MDA)
Gut permeability and health: Inflammatory biomarkers | 0 and 12 weeks
  Change from baseline at week 12: Gut inflammatory biomarkers fecal calprotectin and myeloperoxidase
Biomarkers of inflammation | 0 and 12 weeks
  Change from baseline at week 12: Plasma inflammatory markers (ex. CRP and IL-6)

SECONDARY OUTCOMES:
Urolithin concentrations | 0 and 12 weeks
  Change from baseline at week 12: urolithin A and urolithin B concentrations in urine
Blood pressure | 0 and 12 weeks
  Change from baseline at week 12: systolic and diastolic blood pressure
Weight | 0 and 12 weeks
  Change from baseline at week 12: weight

CONTACTS AND LOCATIONS:
Overall Officials: Emily Ho, PhD, Principal Investigator — Oregon State University
Locations (1):
- Oregon State University, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers without IRB approval.

REFERENCES:
- See also: This website provides detailed study information for potential participants as well as an online screening survey to assess potential eligibility. Additionally, 2 in-person screening visits follow the online screening survey to assess eligibility. — https://lpi.pub/WalnutStudy